CLINICAL TRIAL: NCT07254585
Title: An Open-label, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of SYS6010 Combined With Enlonstobart in the Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: SYS6010 Combined With Enlonstobart In Recurrent Or Metastatic Head And Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-018
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6010 combined with enlonstobart group (Experimental): SYS6010 injection and enlonstobart injection will be administrated on a 14-day cycle
  Interventions: Drug: SYS6010 injection; Drug: Enlonstobart injection
- Enlonstobart group (Experimental): Enlonstobart injection will be administrated on a 14-day cycle
  Interventions: Drug: Enlonstobart injection

INTERVENTIONS:
Drug: SYS6010 injection — SYS6010will be administrated on a 14-day cycle
  Arms: SYS6010 combined with enlonstobart group
Drug: Enlonstobart injection — Enlonstobart is a recombinant human anti-PD-1 monoclonal antibody
  Other Names: Enlonstobart will be administrated on a 14-day cycle

SUMMARY:
This study is a n open-label, multi-center, phase II study to evaluate the efficacy and safety of SYS6010 combined with Enlonstobart in the recurrent or metastatic head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 (inclusive) years old, male or females;
2. Participants with histologically confirmed recurrent or metastatic head and neck squamous cell carcinoma who are not suitable for radical surgery or concurrent chemoradiotherapy.
3. For SYS6010 combined with Enlonstobart group: Participants who have not previously received systemic anti-tumor treatment. If participants have received neoadjuvant or adjuvant therapy (or combination targeted therapy), they are eligible if disease progression occurs at least 6 months after the last administration.
4. For Enlonstobart group: Participants who have not previously received immunotherapy are included. For participants who have not previously undergone systemic antitumor treatment, baseline PD-L1 positivity (CPS≥1) must be confirmed by the central laboratory; for participants who have previously received systemic antitumor treatment, there is no restriction on baseline PD-L1 expression.
5. At least one measurable lesion confirmed by CT or MRI scan according to RECIST v1.1 criteria
6. ECOG performance status of 0-1;
7. Life expectancy ≥ 3 months;
8. Major organ function must meet the criteria within 7 days prior to the first dose of the study intervention
9. Women of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose. Participants must agree to use effective contraception from the time of signing the informed consent form until 7 months after the last dose; during this period, women should not be breastfeeding, and men should avoid donating sperm;
10. Voluntarily participate in this clinical study, understand the study procedures, and be able to sign a written informed consent form.

Exclusion Criteria:

1. The primary sites include the nasopharynx, salivary glands, sinuses, skin, or squamous cell carcinoma of unknown primary origin; Histologically or cytologically confirmed combined neuroendocrine carcinoma, mesenchymal tumors or carcinosarcoma.
2. Patients with meningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or active CNS metastasis. Patients with supratentorial and/or cerebellar metastasis (i.e., without mesencephalon, pons, or medulla involvement) who have received local treatment, have achieved stability for at least 2 weeks prior to the first dose of the study intervention (imaging shows no new brain metastasis or enlargement of existing brain metastasis, and all neurologic symptoms have stabilized or returned to normal), and do not require corticosteroid therapy or are receiving prednisone at a daily dose of ≤10 mg or equivalent doses of other corticosteroids, can participate in the study;
3. Patients with a history of other malignant tumors within 3 years prior to the first dose of the study intervention, except for the following conditions: cured skin basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, and cervical carcinoma in situ, etc.;
4. Patients who are known to be allergic to any component of SYS6010, Enlonstobart or to humanized monoclonal antibody products;
5. AEs caused by prior anti-tumor treatment have not recovered to ≤ Grade 1 (excluding Grade 2 alopecia, peripheral neurotoxicity, and other toxicities judged by the investigator to have no safety risk) according to NCI-CTCAE v5.0;
6. Previously received systemic anti-tumor therapy for locally advanced or metastatic non-squamous NSCLC other than EGFR TKI; patients who have previously received adjuvant/neoadjuvant chemotherapy and experienced disease progression more than 12 months after the end of treatment are allowed to be included;
7. Patients who have not met the corresponding washout period requirements for the medications or treatments should be excluded:
8. History of severe cardiovascular or cerebrovascular disease within 6 months prior to the first dose of the study intervention
9. Imaging examination suggests tumor invasion of the cervical, thoracic, and abdominal great vessels;
10. Patients who have a history of ILD/non-infectious pneumonitis treated with corticosteroids in the past, currently have ILD/non-infectious pneumonitis, for whom imaging examinations at screening cannot rule out ILD/non-infectious pneumonitis, or whose pulmonary function test indicates severe ventilatory dysfunction and/or decreased diffusion capacity;
11. Presence of severe infections within 4 weeks prior to the first dose of the study intervention, including but not limited to bacteraemia requiring hospitalisation, severe pneumonia, active pulmonary tuberculosis infection, etc.; presence of active infections requiring systemic antibiotics within 2 weeks prior to the first dose of the study intervention;
12. Previous interruption of EGFR-targeted therapy for ≥1 month or permanent discontinuation due to skin toxicity, or currently have skin diseases requiring oral or intravenous medication;
13. Participants with active autoimmune diseases or a history of autoimmune diseases (such as ulcerative colitis or Crohn's disease) are excluded, but participants with the following conditions are allowed to proceed to further enrollment screening: well-controlled type 1 diabetes and hypothyroidism that is well-controlled with only hormone replacement therapy.
14. Pleural effusion or pericardial effusion requiring clinical intervention within 2 weeks prior to the first dose;
15. Active HBV or HCV infection (hepatitis B surface antigen and/or hepatitis B core antibody positive and HBV DNA copies ≥ 1×104 copies/mL or ≥ 2000 IU/mL, HCV antibody positive and HCV RNA above the lower limit of detection of the analytical procedure). Note: For HBsAg-positive patients, it is recommended to start antiviral therapy before the first dose of the study intervention, nucleoside analogues are recommended, such as entecavir, tenofovir disoproxil;
16. History of immunodeficiency (including positive HIV test, other acquired or congenital immunodeficiency diseases), history of allogeneic stem cell or organ transplant;
17. Other conditions that the investigator deems unsuitable for participation in this clinical study (such as mental disorders, macular cystoid oedema, severe corneal disorders, uncontrolled or poorly controlled hypertension and diabetes mellitus)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) assessed by investigator | 1 year
Incidences of Adverse Events and Serious Adverse Events | 1 year

SECONDARY OUTCOMES:
Progression Free Survival(PFS) and Overall survival(OS) | 1.5 years
Immunogenicity of SYS6010 and Enlonstobart | 1 year
The plasma concentration of SYS6010 and Enlonstobart | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital Affiliated To Tongji University, Shanghai, Shanghai Municipality, China